CLINICAL TRIAL: NCT06834997
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Groups Study to Explore The Safety And Therapeutic Potential Of Cannabinoids As An Adjunct For Reducing Pain (Carp)- TCH
Brief Title: Dronabinol As an Adjunct for Reducing Pain (DARP)-Texas Children's Hospital
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Christopher D. Verrico, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-56181
Record Dates: First submitted 2025-02-10; First posted 2025-02-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-02

CONDITIONS: Endometriosis; Endometriosis Related Pain; Endometriosis, Pain
Keywords: Endometriosis Related Pain; Endometriosis
MeSH Terms: conditions — Endometriosis; Pain | interventions — Dronabinol

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled, Parallel Groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dronabinol (Experimental): Dronabinol capsules, over-encapsulated with filler to match the appearance of the placebo capsule, up to 15 mg, twice per day for 8 weeks.
  Interventions: Drug: Dronabinol Capsules
- Placebo (Placebo Comparator): Capsules with placebo (i.e., cellulose filler), twice per day for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dronabinol Capsules — Eligible subjects will be randomized (2:1) to dronabinol or placebo, administered orally. The dose of dronabinol will be titrated such that on Day 1, subjects will take 2.5 mg, twice. On subsequent days patients may gradually increase the total number of doses, by one dose each day, as needed and tolerated until either the optimal dose is achieved, or the dose reaches 30 mg THC per day.
  Other Names: Marinol; delta-9-tetrahydrocannabinol
  Arms: Dronabinol
Drug: Placebo — Matching placebo will be prepared and administered in the same manner as the active medication. Titration will occur in a masked fashion such that individuals assigned to placebo undergo a similar perceived titration process.
  Arms: Placebo

SUMMARY:
This exploratory, proof-of-concept study is a double-blind (participants and investigators will be blinded), placebo-controlled, randomized, two-arm clinical trial of Marinol [dronabinol, synthetic Δ9-tetrahydrocannabinol (THC)] for e endometriosis-associated chronic pelvic pain (endo-CPP) with a 2:1 allocation ratio. Up to 75 subjects will be enrolled in this pilot study and randomized to receive doses of THC (up to 30 mg/day), orally, over 8 weeks. This study will be conducted at a single site; it does not include any stratifications, and there is no interim analysis planned. Notably, the goal is to determine whether there is enough evidence of the safety of THC to support the development of later-phase clinical trials. Thus, detailed developmental plans are contingent on the outcomes of this study.

DETAILED DESCRIPTION:
Endometriosis is a progressive, chronic inflammatory disorder that affects approximately 10% of women of reproductive age, with up to 70% to 90% of patients experiencing pelvic pain symptoms, thereby reducing their quality of life, and decreasing labor productivity. Current standard treatments for endometriosis-associated chronic pelvic pain (endo-CPP) include progestin-based hormonal treatments, such as combined oral contraceptive (OC) pills, gonadotropin-releasing hormone (GnRH) analogs, and laparoscopic surgeries. However, endo-CPP often persists even after laparoscopic excision of endometriosis lesions, indicating that controlling disease progression does not necessarily lead to pain relief. As pain is an important factor in endometriosis, optimal analgesia should be sought, which, to date, has primarily been treated with non-steroidal anti-inflammatory drugs (NSAIDs), metamizole, or, in extreme cases, opioids. However, the response to NSAIDs is often ineffective. Additionally, NSAIDs are associated with a higher risk of gastrointestinal bleeding. As for metamizole, agranulocytosis is the most notorious adverse event, along with metamizole-associated hepatotoxicity. Although opioids are generally not recommended for pain relief in women with endometriosis, opioid prescriptions have been identified for women diagnosed with endometriosis within the past year in the United States (As-Sanie S, 2021). Patients undergoing robotic surgery for endometriosis use over two times as many opioids postoperatively as patients without endometriosis and experience higher perceived postoperative pain. Women with endometriosis have a four-fold greater risk of chronic opioid use compared to those without endometriosis. Opioids are highly addictive, and the use of both synthetic and natural opioids can quickly result in dependence, which includes physical and/or psychological dependence, as well as opioid use disorder. Side effects of opioid medications are generally dose-dependent and include constipation, miosis, sedation, and respiratory depression. However, the efficacy of THC in endo-CPP remains uncertain.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Ability to take oral medication per protocol.
4. Female, aged 18-64 years.
5. Females aged ≥ 18 years clinically diagnosed with endometriosis meeting one of the following criteria: a. Patients with previous surgical confirmation of endometriosis and a high suspicion of recurrence b. Patients with imaging (MRI or ultrasonography) findings highly suggestive of endometriosis and confirmed after surgery.
6. Has chronic endometriosis pain that has persisted at least 3 months and has resulted in pain as determined by the Endometriosis Health Profile Questionnaire (EHP-30).
7. For females of reproductive potential: currently practicing an effective form of two types of birth control, which are defined as those, alone or in combination, that result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly, for at least 1 month prior to screening and agrees to use such a method during study participation and for an additional 4 weeks after the end of study medication administration unless she is surgically sterile, partner is surgically sterile, or she is postmenopausal (one year): a. contraceptive sponge, b. patch, c. double barrier (diaphragm/spermicidal or condom/spermicidal), d. intrauterine contraceptive system, e etonogestrel implant, f. medroxyprogesterone acetate contraceptive injection, g. complete abstinence from sexual intercourse, and/or hormonal vaginal contraceptive ring.
8. Patients using oral contraceptives, vaginal ring for contraception and/or management of endometriosis, can be included if both they and their primary provider agree to stopping their medication and transitioning to dronabinol (THC) as the primary treatment of endometriosis throughout the study period
9. Agreement to adhere to Lifestyle Considerations (see section 5.3) throughout study duration.
10. On a stable pain treatment (pharmacological or otherwise) for ≥3 months at the time of the screening and agree to refrain from adding new analgesic medications or increasing their current dose of analgesic medications for the duration of the study.
11. Due to the inability to translate patient facing documents into various languages the investigators will only recruit English speaking participants

Exclusion Criteria:

1. Current and unwilling to stop use of cannabis/marijuana and any other cannabinoids (CBD), including over the counter CBD products.
2. Known allergic reactions to cannabis, CBD, THC, or components of the study interventions.
3. Have Blood Urea Nitrogen or Creatinine levels outside the normal range, or other clinically significant laboratory abnormalities
4. Current use of automated external defibrillator (AED)
5. Chronic daily opioid use and any chronic pain or frequently reoccurring pain condition, other than endometriosis, that is treated with opioids for > 14 days per month
6. Women with a BMI > 35 kg/m2
7. Current use of barbiturates, benzodiazepines, ethanol, lithium, buspirone, muscle relaxants which in the opinion of the P.I. and/or the admitting clinician would preclude the safe and/or successful completion of the study.
8. Current use of amphetamines, other sympathomimetic agents, atropine, amoxapine, scopolamine, antihistamines, other anticholinergic agents, amitriptyline, or desipramine, within 3 months of randomization
9. Treatment with another investigational drug or other intervention within 3 months of the screening visit.
10. Pregnancy, plans to become pregnant, or lactation.
11. Any interventional pain procedures within 6 weeks prior to screening or at any point during study enrollment.
12. Surgical intervention or introduction/increased dose of an opioid or analgesic regimen at any point during study enrollment
13. Implanted spinal cord or dorsal root ganglion stimulator for pain treatment.
14. Meets DSM-V criteria for a current major psychiatric illness, such as bipolar disorder, or psychosis which in the opinion of the P.I. and/or the admitting clinician would preclude the safe and/or successful completion of the study.
15. Have a history of substance abuse or dependence which in the opinion of the P.I. and/or the admitting clinician would preclude the safe and/or successful completion of the study.
16. Have an increased risk of suicide that necessitates inpatient treatment or warrants therapy excluded by the protocol, and/or current suicidal plan, per investigator clinical judgement, based on interview and defined on the Columbia Suicidality Severity Rating Scale (C-SSRS).
17. Have a history of seizures which in the opinion of the P.I. and/or the admitting clinician would preclude the safe and/or successful completion of the study.
18. Have uncontrolled renal, hepatic, or other systemic disorders that in the opinion of the clinician may jeopardize the patient's safe participation in this study.
19. Have a history of cardiac disorders which in the opinion of the P.I. and/or the admitting clinician would preclude the safe and/or successful completion of the study.
20. Myocardial infarction or stroke in the previous 6 months.
21. Resting heart rate of > 120 or Systolic blood pressure > 140 mm Hg, or diastolic blood pressure > 90 mm Hg.
22. Any uncontrolled communicable disease (e.g., HIV/AIDS, tuberculosis, COVID, etc.) which in the opinion of the P.I. and/or the admitting clinician would preclude the safe and/or successful completion of the study.
23. Have any other illness, condition, or use of medications, which in the opinion of the P.I. and/or the admitting clinician would preclude the safe and/or successful completion of the study.
24. Have ECG abnormalities at screening including but not limited to bradycardia (less than 55 beats per minute); prolonged QTc interval (greater than 450 msec); Wolff-Parkinson White syndrome; wide complex tachycardia; 2nd degree, Mobitz type II heart block; 3rd degree heart block; left or right bundle branch block.
25. Have chronic alcohol use (defined as greater then 3 drinks per day, averaged over one week)
26. Known history of or suspected breast cancer on screening physical exam
27. Current use of a progestin-containing contraceptive implant

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Baseline to 8-weeks
  For change in pain intensity from baseline to 8-weeks, the investigators will estimate the mean within each arm using the The Endometriosis Health Profile Questionnaire (EHP-30). 30 point scale ranging from 0 (Never) to 5 (Always).
Safety Analysis | Baseline to 8-weeks
  AEs will be coded using the most recent version of the Medical Dictionary of Regulatory Activities (MedDRA) preferred terms and will be grouped by system, organ, and class (SOC) designation. The severity, frequency, and relationship of AEs to investigational product will be presented by preferred term by SOC grouping. Listings of each individual AE including start date, stop date, severity, relationship, outcome, and duration will be provided.

SECONDARY OUTCOMES:
Analgesic Use Log | Baseline to 8-weeks
  Analgesic Use Change in Analgesic Use Log scores Day 1 to 56 Secondary analyses will use proper tests and appropriate statistical methods at a significance level of 0.05 (2-sided).
Patient-Reported Outcomes Measurement Information System (PROMIS-29) | Baseline to 8-weeks
  The severity of pain will be assessed by the validated scale within the Patient-Reported Outcomes Measurement Information System (PROMIS) is a 29-item profile instrument that can be used to assess seven subscales of health quality of life (QOL) for each of 8 domains-this outcome measure reports one of the 7 domains, anxiety: Physical Function, Anxiety, Depression, Fatigue, Sleep Disturbance, Ability to Participate in Social Roles and Activities, Pain Interference, and Pain Intensity. Responses rage from 5 (Without any difficulty) to 0 (Unable to do) on the Physical Function item, 1 (Never) to 5 (Always) on Anxiety, Depression, Ability to Participate in Social Roles and Activities items, 1 (Not at all) to 5 (Very Much) on the Fatigue, Sleep Disturbance, and Pain Interference items, 0 (No pain) to 10 (Worst Pain Imaginable ) on the Pain Intensity.
Profile of Mood States (POMS questionnaire) | Baseline to 8-weeks
  Changes in POMS . Scale range is 1 to 5 and describes how the participant feels at the time the assessment is administered. Scale of 1, the lowest score, describes a feeling of Not At All right now for the mood and the scale of 5 gives the highest score representing a feeling of Extremely for the mood.
Visual Pain Scale | Baseline to 8-weeks
  The Faces Pain Scale, a visual analogue scale (VAS), is self-report measure of pain intensity on the widely accepted 0-to-10 metric.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Verrico, PhD in Pharmacology, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Hosuton, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fitzcharles MA, Baerwald C, Ablin J, Hauser W. Efficacy, tolerability and safety of cannabinoids in chronic pain associated with rheumatic diseases (fibromyalgia syndrome, back pain, osteoarthritis, rheumatoid arthritis): A systematic review of randomized controlled trials. Schmerz. 2016 Feb;30(1):47-61. doi: 10.1007/s00482-015-0084-3. PMID 26767993